CLINICAL TRIAL: NCT01662336
Title: Real-Life Effectiveness of the Kaletra Adherence Support Assistance (KASA) Program: A Prospective Observational Cohort Study (KASA PMOS)
Brief Title: Real-life Effectiveness of the Kaletra Adherence Support Assistance (KASA) Program
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-566
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: Human Immunodeficiency Virus infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lopinavir/Ritonavir + KASA: Patients were treated according to the standard of care provided by their respective study sites. Treatments with LPV/r and participation in the KASA program were according to the decision of the treating physician and the participant, and were not affected in any way by their decision to participate in the study.
  Interventions: Drug: Lopinavir / ritonavir; Behavioral: Kaletra Adherence Support Assistance Program

INTERVENTIONS:
Drug: Lopinavir / ritonavir — Prescribed according to the product monograph and physician's discretion.
  Other Names: Kaletra®; LPV/r
Behavioral: Kaletra Adherence Support Assistance Program — A customized support network for patients treated with lopinavir / ritonavir that offers individual counseling with an HIV experienced nurse who assists patients with various aspects of their therapy including life-style changes, emotional stress, and adverse events, and may provide access to various healthcare professionals or may offer other types of support such as transportation, exercise, etc.
  Other Names: KASA

SUMMARY:
The overall purpose of the study was to describe the real-life adherence, effectiveness and safety of the Kaletra Adherence Support Assistance (KASA) Program in human immunodeficiency virus (HIV)-positive patients who were receiving treatment with lopinavir / ritonavir (LPV/r; Kaletra®) in Canada.

DETAILED DESCRIPTION:
The Kaletra Adherence Support Assistance (KASA) Program is a customized support network that has been offered to patients treated with lopinavir / ritonavir (LPV/r; Kaletra®). KASA offers individual counseling with an HIV experienced nurse who assists patients with various aspects of their therapy including life-style changes, emotional stress, and adverse events. Patients enrolled in KASA may also have access to various healthcare professionals (dietician, social worker, psychologist, etc.) or may be offered other types of support (transportation, exercise, etc.), which may help improve their quality of life as well as adherence or compliance while taking LPV/r.

This was a 12-month, multi-center, Canadian Post Marketing Observational Study utilizing a prospective single cohort design. All treatments including participation in the KASA program were according to the decision of the treating physician and the patients and were not affected in any way by their decision to participate in the study. Follow-up was for 12 months at an interval of every six months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is HIV-positive
* On treatment with LPV/r or currently initiated on treatment with LPV/r.
* Has provided written informed consent allowing the use of their data for the study and providing permission for contact by the study personnel.
* Willing to be enrolled in the Kaletra Adherence Support Assistance (KASA) program.
* Prescribed LPV/r as part of his/her treatment by the treating physician.

Exclusion Criteria:

* Not willing to sign an informed consent.
* In the opinion of the treating physician is unlikely to be available for the 12-month follow-up duration of the study.
* Is currently participating in a clinical trial of an investigational product.
* Not willing to participate in the KASA program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were enrolled from the offices (at clinic or hospital) of primary care physicians across Canada treating HIV-positive patients.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Pelizon, MD, Study Director — AbbVie Corporation

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the practices of 8 physicians in Canada between 29 June 2012 and 06 August 2015.
Groups:
- Lopinavir/Ritonavir + KASA: Patients were treated according to the standard of care provided by their respective study sites. Treatments with lopinavir / ritonavir (LPV/r; Kaletra®) and participation in the Kaletra Adherence Support Assistance (KASA) program were according to the decision of the treating physician and the participant, and were not affected in any way by their decision to participate in the study.
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir + KASA
Started | 173
Completed Month 6 Visit | 142
Completed Month 12 Visit | 109
Completed | 107
Not Completed | 66
Not completed — Adverse Event | 1
Not completed — No longer on LPV/r | 30
Not completed — Other | 29
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaska | 7
  Asian | 13
  Black | 15
  Hispanic or Latino | 1
  Other | 5
  White | 130
  Missing | 2
Adherence Self-Efficacy Scale (ASES) Scores [Mean (Standard Deviation); unit: units on a scale] — The ASES is a 12 item tool that measures patient's confidence to undertake treatment related activities and behaviors including medication regimen, diet and exercise. Each question is answered on a scale from 0 (cannot do at all) to 10 (certain can do). A summative score ranges from 0 to 120, with higher scores indicating higher treatment self-efficacy. The 12 items converge to two subscales measuring adherence integration and adherence perseverance. The adherence integration subscale score ranges from 0 to 90 and the adherence perseverance subscale score ranges from 0 to 30. Population: Intent-to-treat population included all enrolled participants who received at least 1 dose of lopinavir/ritonavir; data are reported for participants with non-missing data at baseline.
  units on a scale
    Adherence Summative Score: number analyzed (Participants) | 164
    Adherence Summative Score | 102.5 (17.3)
    Adherence Integration Subscale Score: number analyzed (Participants) | 168
    Adherence Integration Subscale Score | 77.1 (13.2)
    Adherence Perseverance Subscale Score: number analyzed (Participants) | 164
    Adherence Perseverance Subscale Score | 25.0 (5.0)
Health Status Assessment (HSA) [Mean (Standard Deviation); unit: units on a scale] — Quality of life (QoL) was measured by the QoL 601-2 survey, the Health Status Assessment (HSA), a brief, comprehensive measure of health-related QoL used extensively in patients with human immunodeficiency virus / acquired immune deficiency syndrome (HIV/AIDS). The survey includes 21 items assessing 8 domains of health-related QoL including physical functioning, role functioning, social functioning, cognitive functioning, pain, energy / fatigue, mental health, and general health perception. Each domain score ranges from 0 to 100 with higher scores indicating higher quality of life. Population: Intent-to-treat population with non-missing data at baseline
  units on a scale
    General Health Perception: number analyzed (Participants) | 166
    General Health Perception | 58.2 (23.2)
    Physical Functioning: number analyzed (Participants) | 169
    Physical Functioning | 67.8 (26.2)
    Role Functioning: number analyzed (Participants) | 168
    Role Functioning | 68.3 (29.5)
    Social Functioning: number analyzed (Participants) | 165
    Social Functioning | 67.8 (26.4)
    Cognitive Functioning: number analyzed (Participants) | 167
    Cognitive Functioning | 64.0 (24.3)
    Pain: number analyzed (Participants) | 167
    Pain | 64.4 (24.8)
    Mental Health: number analyzed (Participants) | 168
    Mental Health | 61.3 (22.6)
    Energy/ Fatigue: number analyzed (Participants) | 168
    Energy/ Fatigue | 54.8 (21.6)
Patient Perception of Stress [Mean (Standard Deviation); unit: units on a scale] — Perception of stress was measured by the Perceived Stress Scale (PSS), a 10-item questionnaire that assesses the degree to which the participant considered situations as stressful. The PSS score ranges from 0 to 40, with higher scores indicating higher levels of perceived stress. Population: Intent-to-treat population with non-missing data at baseline
  units on a scale
    number analyzed (Participants) | 166
    (all) | 16.3 (7.5)
Psychological Well-being [Mean (Standard Deviation); unit: units on a scale] — Psychological well-being was measured by the Center for Epidemiologic Studies Depression scale (CES-D), a 20-item questionnaire assessing the presence of depressive state during the previous week. The possible range of scores is 0 to 60, with higher scores indicating the presence of more symptomatology. Population: Intent-to-treat population with non-missing data at baseline
  units on a scale
    number analyzed (Participants) | 169
    (all) | 18.4 (11.6)
Coping Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — Coping self-efficacy was measured by the Coping Self-Efficacy Scale (CSE), a 26-item questionnaire that measures perceived self-efficacy in coping with daily psychological challenges. A summative score ranging from 0 to 260 was calculated, with higher scores indicating higher coping self-efficacy. Population: Intent-to-treat population with non-missing data at baseline
  units on a scale
    number analyzed (Participants) | 168
    (all) | 187.0 (42.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Adherent to Treatment at Month 6
Description: Adherence was assessed by the Adherence Self-Efficacy Scale (ASES). The ASES is a 12 item tool that measures the patient's confidence to undertake treatment related activities and behaviors including medication regimen, diet and exercise. Each question is answered on a scale from 0 (cannot do at all) to 10 (certain can do). A summative score ranging from 0 to 120 was calculated, with higher scores indicating higher treatment self-efficacy. A participant was considered to have maintained adherence if the change in the ASES summative score at month 6 relative to Baseline was greater than or equal to zero. Participants who discontinued from the study or were lost to follow-up were considered non-adherent.
Time Frame: Baseline and 6 months
Population: The intent-to treat population included all enrolled participants who received at least 1 dose of lopinavir/ritonavir; participants with missing information on the absolute change in the ASES summative score who were not discontinued from the study or lost to follow-up were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 157
percentage of participants | 43.3 [35.9 to 50.7]

2. Secondary Outcome: Change From Baseline in Adherence Summative Score at Months 6 and 12
Description: Adherence was assessed by the Adherence Self-Efficacy Scale (ASES). The ASES is a 12-item tool that measures the participant's confidence to undertake treatment-related activities and behaviors including medication regimen, diet and exercise. Each question was answered on a scale from 0 (cannot do at all) to 10 (certain can do). A summative score ranging from 0 to 120 was calculated, with higher scores indicating higher treatment self-efficacy.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 164
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 126
  Change from Baseline to Month 6 | -1.2 (16.9)
  Change from Baseline to Month 12: number analyzed (Participants) | 93
  Change from Baseline to Month 12 | -5.1 (21.1)

3. Secondary Outcome: Change From Baseline in Adherence Integration Subscale Score at Months 6 and 12
Description: Adherence was assessed by the Adherence Self-Efficacy Scale (ASES). The ASES is a 12-item tool that measures the patient's confidence to undertake treatment-related activities and behaviors including medication regimen, diet and exercise. Each question was answered on a scale from 0 (cannot do at all) to 10 (certain can do).
  The 12 items converge to two subscales measuring adherence integration and adherence perseverance. The adherence integration subscale score ranges from 0 to 90, with higher scores indicating higher treatment self-efficacy.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 168
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 130
  Change from Baseline to Month 6 | -0.7 (13.1)
  Change from Baseline to Month 12: number analyzed (Participants) | 97
  Change from Baseline to Month 12 | -3.6 (15.8)

4. Secondary Outcome: Change From Baseline in Adherence Perseverance Subscale Score at Months 6 and 12
Description: Adherence was assessed by the Adherence Self-Efficacy Scale (ASES). The ASES is a 12-item tool that measures the patient's confidence to undertake treatment-related activities and behaviors including medication regimen, diet and exercise. Each question was answered on a scale from 0 (cannot do at all) to 10 (certain can do). The 12 items converge to two subscales measuring adherence integration and adherence perseverance. The adherence perseverance subscale score ranges from 0 to 30, with higher scores indicating higher treatment self-efficacy.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 164
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 126
  Change from Baseline to Month 6 | -0.1 (4.9)
  Change from Baseline to Month 12: number analyzed (Participants) | 94
  Change from Baseline to Month 12 | -1.0 (6.2)

5. Secondary Outcome: Percentage of Participants Adherent to Treatment at Month 12
Description: Adherence was assessed by the Adherence Self-Efficacy Scale (ASES). The ASES is a 12 item tool that measures the patient's confidence to undertake treatment related activities and behaviors including medication regimen, diet and exercise. Each question was answered on a scale from 0 (cannot do at all) to 10 (certain can do). A summative score ranging from 0 to 120 was calculated, with higher scores indicating higher treatment self-efficacy. A participant was considered to have maintained adherence if the change in the ASES summative score at month 12 was greater than or equal to zero. Participants who discontinued from the study or were lost to follow-up were considered non-adherent.
Time Frame: Baseline and 12 months
Population: The intent-to treat population; participants with missing information on the absolute change in the ASES summative score who were not discontinued from the study or lost to follow-up were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 159
percentage of participants | 30.2 [23.3 to 37.0]

6. Secondary Outcome: Change From Baseline in Health-related Quality of Life General Health Perception Domain Score
Description: Participant quality of life (QoL) was measured by the QoL 601-2 survey, the Health Status Assessment (HSA). This survey is a brief, comprehensive measure of health-related QoL used extensively in patients with human immunodeficiency virus / acquired immune deficiency syndrome (HIV/AIDS). The instrument includes 21 items assessing 8 domains of health-related quality of life including physical functioning, role functioning, social functioning, cognitive functioning, pain, energy / fatigue, mental health, and general health perception. Each domain score ranges from 0 to 100 with higher scores indicating higher quality of life.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 166
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 128
  Change from Baseline to Month 6 | -1.0 (17.6)
  Change from Baseline to Month 12: number analyzed (Participants) | 97
  Change from Baseline to Month 12 | 1.5 (17.7)

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life Physical Functioning Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 169
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 132
  Change from Baseline to Month 6 | 0.0 (21.8)
  Change from Baseline to Month 12: number analyzed (Participants) | 99
  Change from Baseline to Month 12 | 0.1 (22.2)

8. Secondary Outcome: Change From Baseline in Health-related Quality of Life Role Functioning Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 168
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 131
  Change from Baseline to Month 6 | -0.4 (26.5)
  Change from Baseline to Month 12: number analyzed (Participants) | 99
  Change from Baseline to Month 12 | 0.8 (27.1)

9. Secondary Outcome: Change From Baseline in Health-related Quality of Life Social Functioning Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 165
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 129
  Change from Baseline to Month 6 | 0.4 (20.3)
  Change from Baseline to Month 12: number analyzed (Participants) | 96
  Change from Baseline to Month 12 | 2.9 (23.5)

10. Secondary Outcome: Change From Baseline in Health-related Quality of Life Cognitive Functioning Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 167
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 130
  Change from Baseline to Month 6 | 1.2 (18.3)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | 4.7 (18.3)

11. Secondary Outcome: Change From Baseline in Health-related Quality of Life Pain Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 167
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 130
  Change from Baseline to Month 6 | -0.3 (17.7)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | -1.0 (19.5)

12. Secondary Outcome: Change From Baseline in Health-related Quality of Life Mental Health Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 168
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 131
  Change from Baseline to Month 6 | -3.0 (20.5)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | -1.4 (16.5)

13. Secondary Outcome: Change From Baseline in Health-related Quality of Life Energy/ Fatigue Domain Score
Description: as for outcome 6
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 168
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 131
  Change from Baseline to Month 6 | -2.4 (21.0)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | -0.1 (16.7)

14. Secondary Outcome: Change From Baseline in Patient Perception of Stress
Description: Change in perception of stress was measured by the Perceived Stress Scale (PSS), a 10-item questionnaire that assesses the degree to which the participant considered situations as stressful. The PSS score ranges from 0 to 40, with higher scores indicating higher levels of perceived stress.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 166
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 130
  Change from Baseline to Month 6 | -0.3 (9.3)
  Change from Baseline to Month 12: number analyzed (Participants) | 95
  Change from Baseline to Month 12 | -0.8 (9.1)

15. Secondary Outcome: Change From Baseline in Psychological Well-being
Description: Change in psychological well-being was measured by the Center for Epidemiologic Studies Depression scale (CES-D), a 20-item questionnaire assessing the presence of depressive state during the previous week. The possible range of scores is 0 to 60, with higher scores indicating the presence of more symptomatology.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 169
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 132
  Change from Baseline to Month 6 | 1.7 (10.6)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | 1.0 (10.0)

16. Secondary Outcome: Change From Baseline in Coping Self-Efficacy
Description: Change in coping self-efficacy was measured by the Coping Self-Efficacy Scale (CSE), a 26-item questionnaire that measures perceived self-efficacy in coping with daily psychological challenges. A summative score ranging from 0 to 260 was calculated, with higher scores indicating higher coping self-efficacy.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 168
units on a scale
  Change from Baseline to Month 6: number analyzed (Participants) | 129
  Change from Baseline to Month 6 | 2.4 (64.4)
  Change from Baseline to Month 12: number analyzed (Participants) | 98
  Change from Baseline to Month 12 | 8.1 (54.9)

17. Secondary Outcome: Health Resource Utilization
Description: Health resource utilization (HRU) was measured by a self-administered questionnaire that contained a series of questions aimed at measuring the patient's utilization of healthcare resources and economic impact of the disease.
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 173 | 142 | 109
percentage of participants
  Emergency Room | 8.1 | 8.5 | 5.5
  Admitted to Hospital | 3.5 | 2.8 | 3.7
  Admitted to a Long-Term Care Facility | 0.0 | 0.7 | 0.9
  Visit to a Doctor's Office/ Clinic | 55.5 | 50.7 | 50.5
  Ambulance Service | 2.9 | 1.4 | 1.8
  Physiotherapist/ Rehabilitation | 3.5 | 7.7 | 8.3
  Psychiatrist/ Psychologist/ Counselor | 9.2 | 12.0 | 12.8
  Nursing Services | 12.7 | 14.8 | 11.0
  Specialist | 16.2 | 12.7 | 14.7

18. Secondary Outcome: Viral Load at Each Visit
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at baseline and each time point
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 172
copies/mL
  Baseline | 111.3 (10.1)
  Month 6: number analyzed (Participants) | 136
  Month 6 | 55.7 (3.7)
  Month 12: number analyzed (Participants) | 101
  Month 12 | 47.2 (2.5)

19. Secondary Outcome: Cluster of Differentiation 4 (CD4) Positive Cell Counts at Each Visit
Time Frame: Baseline, Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at each time point
Measure: Mean (Standard Deviation); unit: cells/mm³
Arm/Group | Lopinavir/Ritonavir + KASA
Number analyzed (Participants) | 171
cells/mm³
  Baseline | 547.0 (294.21)
  Month 6: number analyzed (Participants) | 135
  Month 6 | 620.8 (294.88)
  Month 12: number analyzed (Participants) | 100
  Month 12 | 620.2 (301.45)

20. Secondary Outcome: Healthcare Provider Satisfaction
Description: For each participant, healthcare provider (HCP) satisfaction with the KASA program was measured by three questions assessing 1) the overall satisfaction with the KASA program, 2) subjective assessment on whether the KASA program was beneficial in maintaining adherence with HIV treatments, and 3) the likelihood of recommending KASA in the future. The scores for each question ranged from 0 to 100, with higher scores indicating higher satisfaction.
Time Frame: Month 6 and Month 12
Population: Intent-to-treat population with non-missing data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Month 6 | Month 12
Number analyzed (Participants) | 142 | 109
units on a scale
  Overall Satisfaction with KASA Program: number analyzed (Participants) | 142 | 107
  Overall Satisfaction with KASA Program | 74.1 (22.10) | 73.3 (22.16)
  Benefits in Maintaining Treatment Adherence: number analyzed (Participants) | 137 | 107
  Benefits in Maintaining Treatment Adherence | 65.6 (26.38) | 62.7 (25.25)
  Likelihood to Recommend KASA Program in Future: number analyzed (Participants) | 136 | 109
  Likelihood to Recommend KASA Program in Future | 74.7 (21.99) | 70.0 (23.14)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Lopinavir/Ritonavir + KASA
Serious Adverse Events (participants affected / at risk) | 3/173
Other Adverse Events (participants affected / at risk) | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir + KASA (N=173)
Cardiac disorder (Cardiac disorders) | 1
Death (General disorders) | 1
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.